CLINICAL TRIAL: NCT05316493
Title: Weight Management Plus Levonorgestrel Intrauterine System or Megestrol Acetate in Endometrial Atypical Hyperplasia: Multiple Single-arm, Prospective and Open-label Clinical Study
Brief Title: Weight Management Plus LNG-IUS/Megestrol Acetate in Endometrial Atypical Hyperplasia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211036-02
Record Dates: First submitted 2022-03-23; First posted 2022-04-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Atypical Endometrial Hyperplasia; Fertility Issues; Overweight and Obesity
MeSH Terms: conditions — Endometrial Hyperplasia; Infertility; Overweight; Obesity | interventions — Megestrol Acetate; Tablets; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive enhanced lifestyle management to control weight and take LNG-IUS or Megestrol Acetate (MA) for treating EAH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- overweight MA+ILI (Experimental): enrolled overweight (24kg/m2≤BMI<28kg/m2) patients will receive megestrol acetate 160mg po qd plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Megestrol Acetate 160 MG Oral Tablet
- overweight LNG-IUS+ILI (Experimental): enrolled overweight (24kg/m2≤BMI<28kg/m2) patients will be treated with LNG-IUS plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Levonorgestrel-Releasing Intrauterine Contraceptive System (Mirena), 52 Mg
- obese MA+ILI (Experimental): enrolled obese (BMI≥28kg/m2) patients will receive megestrol acetate 160mg po qd plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Megestrol Acetate 160 MG Oral Tablet
- obese LNG-IUS+ILI (Experimental): enrolled obese (BMI≥28kg/m2) patients will be treated with LNG-IUS plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Levonorgestrel-Releasing Intrauterine Contraceptive System (Mirena), 52 Mg

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention (ILI) — dietary guidance, exercise guidance, lifestyle intervention
  Other Names: Weight Management
Drug: Megestrol Acetate 160 MG Oral Tablet — enrolled participants will take Megestrol Acetate 160mg daily
  Other Names: yilizhi
  Arms: obese MA+ILI; overweight MA+ILI
Drug: Levonorgestrel-Releasing Intrauterine Contraceptive System (Mirena), 52 Mg — enrolled patients will be treated with LNG-IUS.
  Other Names: manyuele
  Arms: obese LNG-IUS+ILI; overweight LNG-IUS+ILI

SUMMARY:
To investigate the efficacy of weight management plus levonorgestrel intrauterine system (LNG-IUS) or megestrol acetate (MA) in obese patients with endometrial atypical hyperplasia (EAH) asking for conservative therapy.

DETAILED DESCRIPTION:
Background:

High-efficacy progesterone, such as levonorgestrel intrauterine system (LNG-IUS), megestrol acetate (MA), and medroxyprogesterone acetate(MPA), is the first-line treatment for women with endometrial atypical hyperplasia (EAH) who want to preserve fertility. About 70% to 80% of those patients can achieve complete remission (CR) with a median CR time of about 6 months, but about 20% to 30% of those patients get no response or need longer time to get CR (over one year or even longer).

Overweight or obesity is an independent risk factor for fertility-sparing treatment response and pregnancy outcomes in young females with EAH or early endometrioid cancer (EEC). Evidence showed that obesity can cause lower CR rates and longer time to get CR and lower birth rates in EAH or EEC patients asking for conservative therapy. Weight management has been proved to improve metabolic disorders, ovarian functions, and pregnancy outcomes. Metformin, as a diabetes drug, has been proved to increase CR rates in EAH or EEC patients treated with MA for fertility. Weight management has raised more and more attention and has been proved to benefit metabolic and pregnancy outcomes. Based on previous research and published studies, the hypothesise is that weight management plus progestin therapy may raise CR rates and pregnancy outcomes in young female EAH patients asking for fertility conservation.

Enhanced lifestyle management (diet control, exercise, and daily behavioral guidance) may improve metabolic conditions, increase CR rates and pregnancy outcomes in obese EAH patients who want to preserve fertility. Till now, no similar studies were found, so this study is designed to explore the efficacy of weight control in EAH fertility-sparing patients to provide new evidence for improving conservative treatment.

Objective:

To investigate whether weight management plus LNG-IUS/MA can improve the efficacy of preserving fertility in obese EAH women who want fertility conservation.

Design:

This study is designed according to Simon's Two-Stage Design. Based on BMI and treatment plans, four single-arms are designed. This study is prospective, open-label. EAH Patients requiring conservation treatment with BMI ≥ 24 kg/m2 will be recruited in this study and they will be divided into four arms, the first group recruits overweight (24kg/ m2≤BMI<28kg/m2) patients treated with LNG-IUS, the second group recruits overweight (24kg/ m2≤BMI<28kg/m2) patients treated with MA, the third group recruits obese (BMI≥28kg/m2) patients treated with LNG-IUS, and the last group recruits obese (BMI≥28kg/m2) patients treated with MA. The sample size is calculated based on Simon's Two-Stage Design and previous CR rates. All enrolled patients will receive enhanced lifestyle management to control weight and take LNG-IUS/MA for treating EAH. Hysteroscopic examination, metabolic and inflammatory indicators will be performed every 12 to16 weeks while other indexes will be evaluated every month, including weight, heart rates, blood pressure, body fat tests, and so on. For the progestin efficacy evaluation, CR is defined as the remission of EAH to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypia; no response (NR) is defined as the persistence of the disease, and progressive disease (PD) is defined as disease progression in patients. Two months' maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

Outcomes: Primary outcome is the CR rates of the four arms. Secondary outcomes include pregnancy rates, live birth rates, weight loss, insulin resistance, chronic inflammation indicators, time to achieve CR and recurrence rates, and so on. Safety and side events during the whole trial will be monitored in two years.

ELIGIBILITY:
Inclusion Criteria:

1.18 years≤age≤45years 2.BMI (body mass index) ≥24kg/m2 3.Consent informed and signed 4.Pathologically confirmed as endometrial atypical hyperplasia. Patients with endometrial specimens obtained by endometrial biopsy, diagnostic curettage or hysteroscopy and diagnosed histologically as endometrial atypical hyperplasia. If specimens are from other hospitals, they must be counseled or reconfirmed by the Department of Pathology of the Obstetrics and Gynecology Hospital of Fudan University.

5.Have a strong desire to reproduce and ask for fertility preservation or those who insist on keeping the uterus despite no reproductive requirements.

6.Have good compliance and follow-up conditions, and patients are willing to follow up in Obstetrics and Gynecology Hospital of Fudan University in time.

Exclusion Criteria:

1. Combined with severe medical disease or liver or kidney dysfunction: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level elevates to 3 times or more of the upper limit of normal, kidney dysfunction (creatinine clearance < 30 mL/min)
2. Patients are diagnosed with other malignant tumors of the reproductive system; patients with breast cancer or other hormone-dependent tumors that cannot be used with progesterone.
3. Those who have received high doses of high potency progestin or oral contraceptives within the last 3 months (or those on maintenance medication).
4. Those who require hysterectomy or other methods other than conservative treatment.
5. Known or suspected pregnancy.
6. Those who has contraindications to use progestin.
7. Deep vein thrombosis, stroke, myocardial infarction.
8. Severe joint lesions that prevent walking or movement.
9. untreated or recurrent pelvic inflammatory disease (PID)
10. an untreated or uncontrolled pelvic infection (vaginal, cervical, uterine);
11. Cervical dysplasia
12. Congenital or acquired uterine abnormalities, including uterine fibroid tumors or conditions that affect the shape of the uterus
13. allergic to the LNG-IUS components
14. uterine cavity is too large (average uterine diameter is over 7 cm) or have a history of LNG-IUS falling out.

Notes: the last 6 criteria are only applied for patients with LNG-IUS.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (CR) rates | From date of recruitment until the date of CR, assessed up to 28 weeks.
  The 28-week CR rates will be calculated in four arms

SECONDARY OUTCOMES:
Pregnancy outcomes | up to 2 years after complete response of the last participant
  For participants have a desire for fertility, pregnancies, births and related outcomes will be counted, and the rate of pregnancy will be counted as number of pregnancies/ number of patients trying to fertility in the following period.
Weight change | From date of recruitment, assessed up to 28 weeks.
  The investigators will record body weight every month and calculate its change in kilograms.
Body composition change | From date of recruitment, assessed up to 28 weeks.
  The investigators will detect body composition with InBody machine and calculate changes of the indicated indexes.
Blood pressures change | From date of recruitment, assessed up to 28 weeks.
  Record blood pressures (systolic and diastolic pressures) every 12-16 weeks and count the change during the trial.
Heart rates change | From date of recruitment, assessed up to 28 weeks.
  Record heart rates (beats per minute) every 12-16 weeks and count the change.
Blood glucose change | From date of recruitment, assessed up to 28 weeks.
  Assess fasting glucose levels each 3 to 4 months and calculate changes in mmol/L.
Blood lipids change | From date of recruitment, assessed up to 28 weeks.
  Assess blood lipids levels each 3 to 4 months and calculate changes during the trial.
Insulin resistance change | Baseline，3months and 6months after enrolled.
  Test fasting insulin levels each 3 to 4 months, and count HOMA-IR index (Homeostatic Model Assessment for Insulin Resistance) with fasting insulin and fasting glucose as follow: Insulin (pmol/L)*glucose (mmol/L)/22.5, and compare the HOMA-IR change during the treatment.
Ovarian reserve function | From date of recruitment, assessed up to 28 weeks.
  Detect serum Anti-Mullerian Hormone (AMH) each 3 or 4 months and calculate its change.
Quality of life change | From date of recruitment, assessed up to 28 weeks.
  Collect the questionnaire SF-36 and count scores change through conservative treatment.
Impact of Weight on Quality of Life | From date of recruitment, assessed up to 28 weeks.
  Collect questionnaire IWQOL- LITE and count scores change through conservative treatment.
Physical activities change | From date of recruitment, assessed up to 28 weeks.
  Collect physical activities questionnaire(IPAQ) and compare scores changes through conservative treatment.
Chronic inflammatory index (TNF-α) change | baseline, 3 months and 6 months after treatment.
  The investigators will detect the levels of TNF-α (fmol/ml) in serum and calculate changes through the whole treatment period.
Chronic inflammatory index (IL-1) change | baseline, 3 months and 6 months after treatment.
  The investigators will detect serum index IL-1 in U/ml and calculate changes through the whole treatment period.
Chronic inflammatory index (IL-6) change | baseline, 3 months and 6 months after treatment.
  The investigators will detect serum index IL-6 in U/ml and calculate changes through the whole treatment period.
Time of pathological complete response (CR) | From date of recruitment until the date of CR, assessed up to 2 years.
  Time of histologic regression from EAH to proliferative or secretory endometrium
Incidence of adverse events | From date of recruitment until the date of CR, assessed up to 2 years.
  Adverse events related with MA, LNG-IUS and weight control. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete regression, they will be counted and the number of recurrence will be divided by number of patients followed up, then the investigators can get the relapse rates.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOJUN CHEN, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No